CLINICAL TRIAL: NCT05112783
Title: Compare the Effects of Two Different Endotracheal Tubes on The Secretion and Bleeding Volume of Patients During Intubation to Facilitate Nasotracheal Tube Advancement Into Trachea Under Video-laryngoscope
Brief Title: Nasal Intubation：a Comparison of Different Endotracheal Tubes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20210124
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-07

CONDITIONS: Intubation Complication
Keywords: Endotracheal Tube intubation General Anesthesia (ETGA); nasotracheal tube

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Henan Tuoren Endotracheal Tube group (Experimental): Uses the Henan Tuoren endotracheal tube to assist the nasal tracheal tube passing the nasal cavity, oropharynx and advanced into the trachea
  Interventions: Device: Henan Tuoren Endotracheal Tube
- Smiths Portex Tracheal tubes group (Experimental): Uses the Smiths Portex endotracheal tube to assist the nasal tracheal tube passing the nasal cavity, oropharynx and advanced into the trachea
  Interventions: Device: Smiths Portex Tracheal Tubes

INTERVENTIONS:
Device: Henan Tuoren Endotracheal Tube — The endotracheal tube is used under the direct view of the electronic imaging laryngoscope.
  Arms: Henan Tuoren Endotracheal Tube group
Device: Smiths Portex Tracheal Tubes — The endotracheal tube is used under the direct view of the electronic imaging laryngoscope.
  Arms: Smiths Portex Tracheal tubes group

SUMMARY:
Either uses two different endotracheal tubes to pass the nasal cavity and to compare the effects on the secretion and bleeding volume of patients during intubation to facilitate nasotracheal tube advancement.

DETAILED DESCRIPTION:
1. Assess the patient's airway before intubation. EKG, blood pressure and SPO2 are monitored during the process.
2. Randomly divided into two groups：Henan Tuoren Endotracheal Tube and Smiths Portex Tracheal tubes.
3. Sedation process：Give Fentanyl 1 ug/kg according to the patient's weight via IV.
4. Give 1.5ml of Lidocaine without Epinephrine and 0.5ml of Lidocaine with Epinephrine to reduce intranasal bleeding.
5. Sedative injection：give Fentanyl 1ug/kg + Thiamylal 5mg/kg + Rocuronium 1mg/kg
6. Anesthesia intubation inducer：Propofol 1mg/kg
7. Intubation
8. Record the bleeding of the oropharyngeal and nasal mucosa、intubation time、Intubation Difficult Scale (IDS score) and number of intubations during intubation.
9. Record oropharynx、nostril and oropharynx bleeding in 3 minutes after completion of intubation.
10. Evaluate the patient's sore throat, hoarse voice, dysphagia, nasal congestion, nose bleeding, and nasal pain every other day.

ELIGIBILITY:
Inclusion Criteria:

* Age:20-65 years
* Undergoing oro-maxillofacial surgery
* Opening mouth > 3 cm
* Denied any systemic disease.
* American Society of Anesthesiologists (ASA) class:I-III

Exclusion Criteria:

* Difficult airway assessed (limited mouth opening, limited neck motion, and thyromental distance < 6cm)
* Previous head and neck surgery history
* Upper abnormal airway diagnosed
* Easily epistaxis
* Both sides nasal cavities obstruction

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
success rate | 10 minutes
  success rate of tube advancement and successful first tube attempt success rate of tube passing through nasal cavity into trachea
time | 10 minutes
  time taken in tube advancement time taken in tube advancement from nostril into trachea in each time interval

SECONDARY OUTCOMES:
post-anesthesia care | 2 days
  post-intubation induced hoarseness and sore throat intubation related hoarseness and sorethroat at post-anesthesia care unit and the next coming morning

CONTACTS AND LOCATIONS:
Overall Officials: Pin-Yang Hu, MD, Principal Investigator — Department of Anesthesiology, Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin District, Taiwan